CLINICAL TRIAL: NCT05714033
Title: A Randomized Trial Comparing a Ventilatory Strategy To Prevent Atelectasis Versus a Lateral Decubitus Strategy During Robotic Bronchoscopy (VESPA vs. LADS Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-0756; NCI-2023-00783 (Other: NCI CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary; Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1, Participants will receive VESAP during the bronchoscopy. Ventilatory Strategy To Prevent Atelectasis versus a Lateral Decubitus Strategy During Robotic Bronchoscopy
  Interventions: Procedure: Ventilatory Strategy To Prevent Atelectasis
- Group 2 (Experimental): Group 2, Participants will receive LADS Lateral Decubitus Strategy During Robotic Bronchoscopy during the bronchoscopy.
  Interventions: Procedure: Lateral Decubitus Strategy (LADS)

INTERVENTIONS:
Procedure: Ventilatory Strategy To Prevent Atelectasis — Given
  Arms: Group 1
Procedure: Lateral Decubitus Strategy (LADS) — Given
  Arms: Group 2

SUMMARY:
To learn if LADS is better than VESPA at preventing atelectasis during a robotic bronchoscopy.

DETAILED DESCRIPTION:
Primary Objective:

To compare the proportion of patients developing target-obscuring atelectasis when using a lateral decubitus strategy (LADS) vs using a ventilatory strategy to prevent atelectasis (VESPA) during robotic bronchoscopy for posteriorly-located peripheral lung lesions.

Secondary Objectives:

* To compare the proportion of patients with atelectasis in the target lobe in VESPA vs. LADS during robotic bronchoscopy.
* To compare the proportion of patients with atelectasis obscuring 100%, 50% or more, and less than 50% of the target during robotic bronchoscopy using LADS vs. VESPA.
* To compare the proportion of patients in whom a biopsy sample was not taken due to atelectasis using LADS vs. VESPA.
* To compare the diagnostic yield using LADS vs. VESPA.
* To compare the proportion of tool in lesion (TIL) using LADS vs. VESPA.
* To compare the diagnostic accuracy (sensitivity and specificity) for malignancy using LADS vs. VESPA.
* To compare the proportion of LADS-induced vs. VESPA-induced complications.
* To compare the proportion of bronchoscopy-induced complications in LADS vs. VESPA.
* To compare the accuracy of 3D-2D image registration using LADS vs. VESPA.
* To compare clinical workflow in robotic bronchoscopy with VESPA and LADS strategies to identify potential improvements in workflow.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥ 18 years old) undergoing diagnostic robotic bronchoscopy for a lung nodule suspicious for malignancy bronchoscopy under general anesthesia.
2. Lung nodules should be up to 3 cm in diameter and located in right or left bronchial segments B2, B6, B9, and B10. Greater than 50% of the volume of the lesion needs to be below a horizontal line traced at the most anterior edge of the corresponding vertebral body.
3. Chest CT performed < 45 days prior to bronchoscopy.
4. Voluntary informed consent to participate in the study.

Exclusion Criteria:

1. Patients with prior lung consolidation, interstitial changes or lung masses (> 3 cm in diameter) as seen on most recent CT
2. Lesions outside of the designated lung areas defined as inclusion criteria.
3. Known pregnancy
4. Vulnerable population
5. Ascites
6. Known diaphragmatic paralysis
7. Smokers or ex-smokers with known or suspected severe air-trapping defined as residual volume > 150% of predicted
8. History of primary or secondary spontaneous pneumothorax
9. Lung bullae > 5 cm
10. Patients with mediastinal or hilar adenopathy with high suspicion for malignancy in whom lymph node sampling is indicated and should occur prior to robotic bronchoscopy of the peripheral lesion.
11. Patient with active COVID pneumonia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2032-09-14 (Estimated); Study Completion 2032-09-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Casal, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Boster JM, Goertzen M, Sarkiss M, Armas Villalba AJ, Bhandarih BS, Song J, Jimenez CA, Sabath BF, Lin J, Grosu HB, Ost DE, Eapen GA, Chintalapani G, Casal RF. Lateral Decubitus Strategy is Superior to Ventilatory Strategy in Preventing Atelectasis From Obscuring Targets During Robotic Bronchoscopy, Leading to Improved Procedural Outcomes (Lateral Decubitus Strategy vs Ventilatory Strategy to Prevent Atelectasis Trial). Chest. 2026 Jan 8:S0012-3692(25)05835-0. doi: 10.1016/j.chest.2025.11.044. Online ahead of print. PMID 41513124
- See also: M D Anderson Cancer Center — http://www.mdanderson.org